CLINICAL TRIAL: NCT00317044
Title: A 6-month Randomized, Double-blind, Parallel-group, Multicentre, Placebo-controlled Phase II Study to Compare Anti-asthmatic Effect and Safety of Esomeprazole (Nexium®) 40 mg Twice Daily or 40 mg Once Daily With Placebo in Adults With Asthma
Brief Title: Safety and Efficacy Study to Determine Anti-Asthmatic Effect of Esomeprazole Magnesium; Nexium Reflux Asthma
Acronym: RELAX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D9618C00001; RELAX
Record Dates: First submitted 2006-04-20; First posted 2006-04-24 (Estimated); Results first posted 2014-06-09 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-05

CONDITIONS: Asthma; GERD
Keywords: Moderate to severe Asthma; Gastroesophageal Reflux Disease; esomeprazole; GERD
MeSH Terms: conditions — Asthma; Gastroesophageal Reflux | interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Esomeprazole 40 mg twice daily (Experimental)
  Interventions: Drug: Esomeprazole
- Esomeprazole 40 mg once daily (Experimental)
  Interventions: Drug: Esomeprazole
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Esomeprazole — Esomeprazole 40 mg twice daily
  Arms: Esomeprazole 40 mg twice daily
Drug: Esomeprazole — Esomeprazole 40 mg once daily
  Arms: Esomeprazole 40 mg once daily
Drug: Placebo — Placebo twice daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether treatment with esomeprazole for 6 months will improve asthma in adult patients with moderate to severe asthma and symptoms of gastroesophageal reflux disease.

ELIGIBILITY:
Inclusion Criteria:

* Adults with diagnosis of asthma since at least 6 months.
* Symptoms of asthma during run-in.
* At least 3 months history and present symptoms of 1 or more of the following: burning feeling behind breastbone, pain behind breastbone, acid taste in the mouth.

Exclusion Criteria:

* Patients with clinically relevant abnormalities.
* Patients with a smoking history of ≥10 pack-year.
* Patients who have had previous surgery on the esophagus or the stomach.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 961 (Actual)
Dates: Start 2006-04; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Nexium Medical Science Director, MD, Study Director — AstraZeneca
Locations (130):
- United States (27):
  - Research Site, Birmingham, Alabama
  - Research Site, Scottsdale, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Fountain Valley, California
  - Research Site, Miami, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Stockbridge, Georgia
  - Research Site, Normal, Illinois
  - Research Site, Overland Park, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Mandeville, Louisiana
  - Research Site, Wheaton, Maryland
  - Research Site, St Louis, Missouri
  - Research Site, Papillion, Nebraska
  - Research Site, Asheville, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Sylvania, Ohio
  - Research Site, Medford, Oregon
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Upland, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Austin, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Kirkland, Washington
  - Research Site, Seattle, Washington
  - Research Site, Greenfield, Wisconsin
- Argentina (9):
  - Research Site, Ciudad de Buenos Aires, Argentina
  - Research Site, Monte Grande, Buenos Aires
  - Research Site, Quilmes, Buenos Aires
  - Research Site, Córdoba, Córdoba Province
  - Research Site, Córdoba, Córdoba, Argentina
  - Research Site, Rosario, Santa Fe Province
  - Research Site, Rosario, Santa Fe, Argentina
  - Research Site, San Miguel de Tucumán, Tucumán, Argentina
  - Research Site, Buenos Aires
- Bulgaria (5):
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Rousse
  - Research Site, Sofia
  - Research Site, Varna
- Canada (11):
  - Research Site, Calgary, Alberta
  - Research Site, Bay Roberts, Newfoundland and Labrador
  - Research Site, Holyrood, Newfoundland and Labrador
  - Research Site, Brampton, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Woodstock, Ontario
  - Research Site, La Malbaie, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- Czechia (9):
  - Research Site, Benesov U Prahy
  - Research Site, Beroun
  - Research Site, Cvikov
  - Research Site, Kladno
  - Research Site, Kolín
  - Research Site, Liberec
  - Research Site, Prague
  - Research Site, Rokycany
  - Research Site, Tábor
- France (9):
  - Research Site, Brest
  - Research Site, Férolles-Attilly
  - Research Site, Grasse
  - Research Site, Grenoble
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Paris
  - Research Site, Saint-Laurent-du-Var
  - Research Site, Villejuif
- Germany (13):
  - Research Site, Bad Wörishofen
  - Research Site, Berlin
  - Research Site, Frankfurt
  - Research Site, Freising
  - Research Site, Gelnhausen
  - Research Site, Gelsenkirchen
  - Research Site, Hamburg
  - Research Site, Landsberg
  - Research Site, Marburg
  - Research Site, Nuremberg
  - Research Site, Potsdam
  - Research Site, Rodgau-dudenhofen
  - Research Site, Wolmirstedt
- Hungary (9):
  - Research Site, Budapest
  - Research Site, Füzesabony
  - Research Site, Gyöngyös
  - Research Site, Győr
  - Research Site, Hódmezővásárhely
  - Research Site, Kaposvár
  - Research Site, Mosonmagyaróvár
  - Research Site, Százhalombatta
  - Research Site, Szombathely
- Italy (11):
  - Research Site, Cagliari, CA
  - Research Site, Crema, CR
  - Research Site, Florence, FI
  - Research Site, Arenzano, GE
  - Research Site, Palermo, PA
  - Research Site, Pisa, PI
  - Research Site, Prato, PO
  - Research Site, Roma, Roma
  - Research Site, Bussolengo, VR
  - Research Site, Verona, VR
  - Research Site, Napoli
- Mexico (5):
  - Research Site, Guadalajara, Jalisco
  - Research Site, Zapopan, Jalisco
  - Research Site, Morelia, Michoacán
  - Research Site, Villahermosa, Tabasco
  - Research Site, México
- Poland (10):
  - Research Site, Bydgoszcz
  - Research Site, Gdynia
  - Research Site, Iława
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Piekary Śląskie
  - Research Site, Skarżysko-Kamienna
  - Research Site, Strzelce Opolskie
  - Research Site, Tarnów
  - Research Site, Zabrze
- Portugal (4):
  - Research Site, Amadora
  - Research Site, Covilha
  - Research Site, Porto
  - Research Site, Vila Nova de Gaia
- Slovakia (7):
  - Research Site, Bratislava
  - Research Site, Košice
  - Research Site, Nové Zámky
  - Research Site, Považská Bystrica
  - Research Site, Prievidza
  - Research Site, Rimavská Sobota
  - Research Site, Trenčín
- Research Site, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Derived] Kiljander TO, Junghard O, Beckman O, Lind T. Effect of esomeprazole 40 mg once or twice daily on asthma: a randomized, placebo-controlled study. Am J Respir Crit Care Med. 2010 May 15;181(10):1042-8. doi: 10.1164/rccm.200910-1537OC. Epub 2010 Jan 28. PMID 20110554
- See also: CSR-D9618C00001.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=442&filename=CSR-D9618C00001.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Four randomized patients were excluded from the ITT analysis due to missing efficacy data (2 patients), no investigational product given (1 patient), and being unblinded by the investigator (1 patient). The patient who received no investigational product was excluded from the safety analysis and is not included in the Baseline Characteristics.
Groups:
- Esomeprazole 40 mg Twice Daily: Nexium 40 mg given as esomeprazole magnesium trihydrate capsules twice daily
- Esomeprazole 40 mg Once Daily: Nexium 40 mg given as esomeprazole magnesium trihydrate capsules once daily
- Placebo: Placebo
Period: Overall Study
Arm/Group | Esomeprazole 40 mg Twice Daily | Esomeprazole 40 mg Once Daily | Placebo
Started | 320 | 313 | 328
Completed | 272 | 273 | 283
Not Completed | 48 | 40 | 45
Not completed — Protocol Violation | 28 | 22 | 20
Not completed — Adverse Event | 4 | 7 | 4
Not completed — Withdrawal by Subject | 10 | 7 | 12
Not completed — Lost to Follow-up | 0 | 2 | 3
Not completed — Multiple Reasons | 6 | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Esomeprazole 40 mg Twice Daily | Esomeprazole 40 mg Once Daily | Placebo | Total
Number analyzed (Participants) | 319 | 313 | 328 | 960
Age, Continuous [Mean (Full Range); unit: Years] | 44.0 [18 to 69] | 45.0 [19 to 70] | 45.0 [18 to 70] | 44.667 [18 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 240.00 | 240.00 | 247.00 | 727
  Male | 79.00 | 73.00 | 81.00 | 233

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Morning Peak Expiratory Flow (mPEF (L/Minute)) From Baseline (Mean of the Last 7 Days in the run-in Period) to Treatment Period (Mean of All Available Data During the Treatment Period).
Description: Peak expiratory flow is defined as the maximum speed of expiration as measured with the Mini-Wright® PEF Meter. Participants must have both baseline and follow up measure to be included in analysis. Results presented as a mean of all available data during the treatment period.
Time Frame: Baseline to 6 months
Measure: Least Squares Mean (Standard Error); unit: L/minute
Arm/Group | Esomeprazole 40 mg Twice Daily | Esomeprazole 40 mg Once Daily | Placebo
Number analyzed (Participants) | 316 | 311 | 327
L/minute | 21.1891 (2.8689) [lower limit 0] | 19.1847 (2.8422) [0 to 0] | 15.6771 (2.8086) [0 to 0]

2. Secondary Outcome: Changes in Average Value From Baseline to Treatment Period in Evening Peak Expiratory Flow (ePEF (L/Minute))
Description: Peak expiratory flow is defined as the maximum speed of expiration as measured with the Mini-Wright® PEF Meter. Participants must have both baseline and follow up measure to be included in analysis. No dispersion measure available.
Time Frame: Baseline to 6 months
Measure: Least Squares Mean (Standard Error); unit: L/minute
Arm/Group | Esomeprazole 40 mg Twice Daily | Esomeprazole 40 mg Once Daily | Placebo
Number analyzed (Participants) | 316 | 311 | 326
L/minute | 21.88 (2.89) | 18.37 (2.87) | 18.55 (2.83)

3. Secondary Outcome: Changes in Average Value From Baseline to Treatment Period in Asthma Symptom Score - Total
Description: Participants must have both baseline and flow up measure to be included in analysis. Each morning and evening, the patient will be asked to record his/her asthma symptoms (sx) in the diary. The asthma sx scores during night- and daytime will be assessed by the patient according to the following scoring system: 0 = no asthma sx; 1 = you are aware of your asthma sx but can easily tolerate the sx; 2 = your asthma sx are causing you enough discomfort to cause problems with normal activities (or with sleep); 3 = you are unable to do your normal activities (or sleep) because of your asthma. The total symptom score is the sum of the night- and daytime scores.
Time Frame: Baseline to 6 months
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Esomeprazole 40 mg Twice Daily | Esomeprazole 40 mg Once Daily | Placebo
Number analyzed (Participants) | 315 | 311 | 326
Scores on a scale | -0.61 (0.05721) | -0.47 (0.05652) | -0.52 (0.05609)

4. Secondary Outcome: Changes in Average Value From Baseline to Treatment Period in Number of Inhalations of Short-acting β2-agonists (SABAs) - Total From Baseline to 6 Months
Description: This is the change in the average number of inhalations from baseline to the end of the study (6 months). Participants must have both baseline and follow up measure to be included in analysis. Treatment mean calculated using the entire treatment period.
Time Frame: Baseline to 6 months
Measure: Least Squares Mean (Standard Error); unit: Inhalations
Arm/Group | Esomeprazole 40 mg Twice Daily | Esomeprazole 40 mg Once Daily | Placebo
Number analyzed (Participants) | 315 | 311 | 326
Inhalations | -0.77 (0.10) [0 to 17] | -0.73 (0.10) [0 to 13] | -0.68 (0.10) [0 to 14]

5. Secondary Outcome: Changes in Average Value From Baseline to Treatment Period in Percentage of Nights With Awakening(s) Due to Asthma
Description: Change in percentage of nights with night-time awakening(s) due to asthma from baseline to the end of the study (6 months). Participants must have both baseline and follow up measure to be included in analysis.
Time Frame: Baseline to 6 months
Measure: Least Squares Mean (Standard Error); unit: Percent of nights
Arm/Group | Esomeprazole 40 mg Twice Daily | Esomeprazole 40 mg Once Daily | Placebo
Number analyzed (Participants) | 316 | 311 | 327
Percent of nights | -0.238 (0.018) | -0.219 (0.018) | -0.223 (0.018)

6. Secondary Outcome: Change in Forced Expiratory Volume in 1 Second (FEV1) From Randomization to Treatment Period.
Description: Description: Changes in forced expiratory volume in 1 second (FEV1) from randomization (Visit 3) to the treatment period considered as mean value at Visits 4-7. Participants must have both baseline and follow up measure to be included in analysis.
Time Frame: From randomization (Visit 3) to visit 7.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Esomeprazole 40 mg Twice Daily | Esomeprazole 40 mg Once Daily | Placebo
Number analyzed (Participants) | 312 | 306 | 324
Liters | 0.09 (0.02) | 0.07 (0.02) | 0.02 (0.02)

7. Secondary Outcome: Number of Patients With Severe Asthma Exacerbations.
Time Frame: Up to 6 months
Measure: Number; unit: Participants
Arm/Group | Esomeprazole 40 mg Twice Daily | Esomeprazole 40 mg Once Daily | Placebo
Number analyzed (Participants) | 318 | 312 | 327
Participants | 33 | 41 | 43

8. Secondary Outcome: Change in Asthma Quality of Life Questionnaire, Standardized Version (AQLQ(S)) Scores From Randomization (Visit 3) to Visit 7
Description: The Asthma Quality of Life Questionnaire, Standardized Version (AQLQ(S))has been developed by and includes 32 questions in 4 domains: activity limitation, symptoms, emotional function, and exposure to environmental stimuli. It is used to measure the physical and emotional impact of the disease in the selected areas of life. Participants must have both baseline and follow up measure to be included in analysis.AQLQ(S) score based on a 7-point scale that ranged from 1 (worst quality of life) to 7 (best quality of life).
Time Frame: From randomization (Visit 3) to Visit 7
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Esomeprazole 40 mg Twice Daily | Esomeprazole 40 mg Once Daily | Placebo
Number analyzed (Participants) | 272 | 275 | 288
Scores on a scale | 0.97 (0.07) | 0.83 (0.07) | 0.55 (0.07)

9. Secondary Outcome: Change in Symptoms of GERD as Measured by Reflux Disease Questionnaire (RDQ) From Randomization (Visit 3) to Visit 7
Description: The RDQ questionnaire is used to assess six GI symptoms during the previous week (a burning feeling behind the breastbone, pain behind the breastbone, a burning feeling in the centre of the stomach, pain in the centre of the stomach, an acid taste in the mouth, unpleasant movement of material upwards from the stomach). Each symptom is given a frequency score on a six-point scale (from 0=did not have to 5=daily) and an intensity score on a six-point scale (from 0=did not have to 5=severe). Three domain scores are calculated by forming averages of the frequency and intensity scores of selected symptoms (heartburn: the first two symptoms; dyspepsia: the next two symptoms; regurgitation: the last two symptoms). The overall GERD score is calculated as the average of the hearburn and dyspepsia domain scores. The GERD score can thus range from 0 to 5.
Time Frame: Randomization (Visit 3) to Visit 7
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Esomeprazole 40 mg Twice Daily | Esomeprazole 40 mg Once Daily | Placebo
Number analyzed (Participants) | 316 | 311 | 327
Scores on a scale | -1.95 (0.07) | -1.91 (0.07) | -1.27 (0.07)

10. Secondary Outcome: Number of Severe Adverse Events
Time Frame: Up to 6 months
Measure: Number; unit: Events
Arm/Group | Esomeprazole 40 mg Twice Daily | Esomeprazole 40 mg Once Daily | Placebo
Number analyzed (Participants) | 316 | 311 | 327
Events | 4 | 5 | 9

11. Secondary Outcome: Changes in Average Value From Baseline to Treatment Period in Asthma Symptom Score - Night
Description: Participants must have both baseline and follow up measure to be included in analysis
Time Frame: Baseline to 6 months
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Esomeprazole 40 mg Twice Daily | Esomeprazole 40 mg Once Daily | Placebo
Number analyzed (Participants) | 316 | 311 | 327
Scores on a scale | -0.31 (0.03) | -0.23 (0.03) | -0.27 (0.03)

12. Secondary Outcome: Changes in Average Value From Baseline to Treatment Period in Asthma Symptom Score - Day
Description: Participants must have both baseline and follow up measure to be included in analysis
Time Frame: Baseline to 6 months
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Esomeprazole 40 mg Twice Daily | Esomeprazole 40 mg Once Daily | Placebo
Number analyzed (Participants) | 316 | 311 | 327
Scores on a scale | -0.30 (0.03) | -0.25 (0.03) | -0.25 (0.03)

13. Secondary Outcome: Changes in Average Value From Baseline to Treatment Period in Number of Inhalations of Short-acting β2-agonists (SABAs) - Night
Description: Participants must have both baseline and follow up measure to be included in analysis
Time Frame: Baseline to 6 months
Measure: Least Squares Mean (Standard Error); unit: Inhalations
Arm/Group | Esomeprazole 40 mg Twice Daily | Esomeprazole 40 mg Once Daily | Placebo
Number analyzed (Participants) | 316 | 311 | 327
Inhalations | -0.30 (0.05) | -0.27 (0.05) | -0.29 (0.04)

ADVERSE EVENTS:
Arm/Group | Esomeprazole 40 mg Twice Daily | Esomeprazole 40 mg Once Daily | Placebo
Serious Adverse Events (participants affected / at risk) | 7/319 | 5/313 | 5/328
Other Adverse Events (participants affected / at risk) | 37/319 | 44/313 | 55/328
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Esomeprazole 40 mg Twice Daily (N=319) | Esomeprazole 40 mg Once Daily (N=313) | Placebo (N=328)
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Cervical Dysplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis Chronic (Hepatobiliary disorders) | 1 | 0 | 0
Chronic Sinusitis (Infections and infestations) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 1 | 0
Migraine With Aura (Nervous system disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Renal Colic (Renal and urinary disorders) | 1 | 0 | 0
Salmonellosis (Infections and infestations) | 1 | 0 | 0
Sinus Polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Small Intestine Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tuberculosis (Infections and infestations) | 1 | 0 | 0
Umbilical Hernia (Gastrointestinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Esomeprazole 40 mg Twice Daily (N=319) | Esomeprazole 40 mg Once Daily (N=313) | Placebo (N=328)
Bronchitis (Infections and infestations) | 11 | 16 | 18
Upper Respiratory Tract Infection (Infections and infestations) | 26 | 28 | 37

LIMITATIONS AND CAVEATS:
Numbers of patients analyzed in each of the Outcome Measures varies due to the amount of qualifying data captured for the patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days